CLINICAL TRIAL: NCT05228899
Title: A Phase I/II Multicenter, Randomized, Double Blinded, Placebo Trial to Evaluate the Safety and Potential Efficacy of Zofin Infused Intravenous (IV) in Patients Experiencing Prolonged COVID-19 Symptoms (Long-Haulers) vs Placebo.
Brief Title: Zofin to Treat COVID-19 Long Haulers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ZEO ScientifiX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 27378
Record Dates: First submitted 2022-02-02; First posted 2022-02-08 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: COVID-19
Keywords: COVID-19 Long Hauler; PASC; Zofin; Exosomes; Extracellular Vesicles
MeSH Terms: conditions — COVID-19 | interventions — amniotic fluid peptide-1, human; Saline Solution

STUDY DESIGN:
Intervention Model Description: This is a phase I/II randomized, double blinded and placebo control. The ratio between groups is 1:1 for total 30 subjects. Each subject will be randomized to receive either treatment or placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Neither the patients nor the researchers know who is getting a placebo and who is getting the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Zofin (Experimental): Group 1 (15 subjects) Fifteen subjects will receive 1 mL of Zofin diluted with 100ml of sterile saline on day 0, day 4 and day 8, containing 2-5 x 10^11 particles/ml intravenously.
  Interventions: Drug: Zofin
- Group 2: Placebo (Placebo Comparator): Group 2 (15 subjects) Fifteen subjects will receive 1mL of placebo diluted with 100ml of sterile saline on day 0, day 4 and day 8, containing sterile saline intravenously.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Zofin — 1mL of Zofin will be administered intravenously, containing 2-5 x 10^11 particles/mL. Zofin will be diluted in 100 mL of sterile saline.
  Other Names: human amniotic fluid
  Arms: Group 1: Zofin
Other: Placebo — 1mL of Placebo (normal saline) will be diluted in 100 mL of sterile saline and administered intravenously.
  Other Names: normal saline
  Arms: Group 2: Placebo

SUMMARY:
The purpose of this study is to assess the safety and potential efficacy of Zofin administered intravenously in subjects experiencing prolonged symptoms (> 6 weeks and < 24 months) of COVID-19.

DETAILED DESCRIPTION:
This is a phase I/II randomized, double blinded and placebo control. COVID-19 Long Haulers

In double blinded and placebo control trial, neither the patients nor the researchers know who is getting a placebo and who is getting the treatment. The ratio between groups is 1:1 for total 30 subjects. Each subject will be randomized to receive either treatment or placebo.

A total of 30 subjects will be enrolled and randomized.

Group 1 (15 subjects) Fifteen subjects will receive 1 mL of Zofin diluted with 100ml of sterile saline on day 0, day 4 and day 8, containing 2-5 x 10^11 particles/ml intravenously.

Group 2 (15 subjects) Fifteen subjects will receive 1mL of placebo diluted with 100ml of sterile saline on day 0, day 4 and day 8, containing sterile saline intravenously.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age > 18 years at the time of signing the informed consent form.
2. Male or female.
3. COVID-19 survivor and had documented SARS-CoV-2 positive (FDA EUA approved RT-PCR or equivalent tests such as FDA EUA approved Rapid Antigen Test which is performed at CLIA certified lab or the readout of the test reviewed and documented by a doctor).
4. Subject experiencing fatigue for over 6 weeks after their positive test result while currently being negative.
5. Subject has not fully recovered from COVID-19 for at least over 6 weeks despite a negative SARS-COV-02 test.
6. Subjects tested positive for anti-SARS-CoV-2 antibodies using FDA EUA approved test.
7. Subject is experiencing the following three symptoms for at least over 6 weeks either continually or intermittently with relapses not experienced pre-illness, that interferes with normal daily activities. Symptoms must be new symptoms i.e., subject didn't have symptoms, and had not sought medical treatment for the symptoms prior to COVID-19:

   * Extreme fatigue - feeling overtired with low energy and a strong desire to sleep but unable to have good sleep.
   * Body aches - muscle soreness or generalized achiness throughout the body.
   * Joint pain - pain in the joints due to inflammation not experienced before illness.
8. Chalder Fatigue Scale Bimodal Score ≥ 4 at the time of Screening.
9. Fatigue Severity Scale (FSS) ≥ 4 at the time of Screening.
10. Fatigue Assessment Scale Score (FAS) ≥ 10.5 at the time of Screening.
11. Beck Depression Inventory (BDI) score <15 at the time of Screening (score of 15 is an exclusion).
12. Investigator(s) has access to medical documentation of previous COVID-19 treatments.
13. Ability of subject to understand and the willingness to sign a written informed consent document.
14. Subjects must be reasonably able to return for multiple follow-up visits.
15. Adequate venous access.
16. For Subjects of Child-Bearing Potential only, willingness to use FDA recommended birth control until 6 months post-treatment. The FDA approved and cleared methods for birth control are listed below:

    * Permanent sterilization
    * Long-acting reversible contraceptives (LARC)
    * Contraceptive injection
    * Short-acting hormonal methods
    * Barrier methods
    * Emergency contraception https://www.fda.gov/consumers/free-publications-women/birthcontrol
17. Any male subject must agree to use contraceptives and not donate sperm during the study.

Exclusion Criteria:

1. Tested positive for SARS-CoV-2 infection at the time of screening (acute infection) which will involve a nasal swab sample or another FDA-approved test.
2. Subjects with a BDI ≥ 15 are excluded.
3. Subjects with homicidal or suicidal ideation are excluded.
4. Subjects with a diagnosis of depression upon entry into the study must have had at least 2-months of treatment (psychotherapy, antidepressive medication, or both) prior to enrollment, be stable on their current treatment regimen, and be followed by a medical provider who is actively treating and managing their depression throughout the study period.
5. Subjects who had recovered fully from COVID-19 and have a new onset of extreme fatigue, body aches, or joint pain that were due to other etiologies, not COVID-19 are excluded.
6. Subjects with serious co-morbidities are excluded. For example:

   * Liver enzymes are >2X ULN;
   * eGFR is <60 ml/min by the CKD- EPI equation;
   * Hb is <11 mg/dL;
   * Platelet count is <100K;
   * Uncontrolled arrhythmias;
   * BP systolic <90 mmHg or >160 mmHg;
   * Pulse is <60 or >100;
   * Respiratory rate is <12 or >25;
   * Abnormal ECG or any signs of active ischemic heart disease;
   * Heart failure of any degree (including NYHA classification Class 1- 4).
7. History of migraines prior to COVID-19 infection.
8. History of neuropathy prior to COVID-19 infection.
9. History of inflammatory and irritable bowel disease prior to COVID-19 infection.
10. History of depression and anxiety disorders prior to COVID-19 infection.
11. History of chronic fatigue syndrome, fibromyalgia, and arthritic disorders prior to COVID-19 infection.
12. Exhibiting signs of moderate or severe chronic respiratory disease (such as COPD, asthma, or pulmonary fibrosis) and history of these illnesses prior to COVID-19 infection.
13. Patient with rheumatologic disorders.
14. History of chronic liver disease or patient showing signs of clinical jaundice at the time of screening.
15. History of severe chronic kidney disease or requiring dialysis.
16. Showing signs of severe pneumonia, acute respiratory distress syndrome (ARDS), or respiratory failure needing mechanical ventilation.
17. Subjects with a history of bleeding disorders or currently on anticoagulation therapy that cannot be stopped prior to infusion which is not related to previous COVID-19 infection.
18. Oxygen-dependent on nasal canula greater than 2-L per minute.
19. Patient with pulse oxygen saturation (SpO2) of <94% on room air.
20. Active or recently treated malignancies.
21. Any unstable condition of clinical significance, e.g., uncontrolled hypertension, unstable angina pectoris, worsening asthma.
22. Hydroxychloroquine, oral or parenteral corticosteroids, immunosuppressants, or immunomodulating agents within 7 days prior to the screening visit.
23. Albuterol as nebulizer for the off-label treatment of COVID-19 within 7 days prior to the screening visit.
24. Be a female who is pregnant, nursing, or of childbearing potential while not practicing effective contraceptive methods. Female subjects must undergo a blood pregnancy test at screening which will be within 72 hours of the IP infusion.
25. Subject has a body mass index (BMI) greater than 42 kg/m2
26. Subject has or had an active infection requiring systemic antibiotics within 12 weeks of enrollment in the study.
27. Inability to perform any of the assessments required for endpoint analysis.
28. Active listing (or expected future listing) for transplant of any organ.
29. Be a solid organ transplant recipient. This does not include prior cell based therapy (>12 months prior to enrollment), bone, skin, ligament, tendon or corneal grafting.
30. Have a history of organ or cell transplant rejection.
31. History of drug abuse (illegal "street" drugs except marijuana, if it is legal to use in states where patient resides), or prescription medications not being used appropriately for a pre-existing medical condition or alcohol abuse (≥ 5 drinks/day for ˃ 3 months), or documented medical, occupational, or legal problems arising from the use of alcohol or drugs within the past 24 months.
32. Patients with untreated HIV infection. However, patients can be enrolled if have been treated for HIV and the test negative for HIV viral load but still test positive for antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
Incidence of Severe Adverse Events | 30 days
  To evaluate the safety of Zofin administered intravenously in subjects experiencing prolonged COVID-19 symptoms. To compare the incidence of grade 3 or 4 or serious adverse events (SAEs) in subjects receiving Zofin compared to placebo:
  * Occurrence of SAEs within 30 days related to the therapy.
  * Life-threatening event (e.g., stroke or non-fatal pulmonary embolism).
  * Event requiring inpatient hospitalization (e.g., for worsening dyspnea).
  * Event resulting in persistent or significant disability/incapacity.
  * Event resulting in death.

SECONDARY OUTCOMES:
Fatigue Severity Score Score | 0, 8,14, 30, 60 days
  The Fatigue Severity Scale (FSS) is a method of evaluating the impact of fatigue.
Daily Diary of COVID-19 Related Symptom | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 21, 28 days
  Changes in daily COVID-19-Related Symptom Severity Score during the treatment phase
COVID-19 Associated Symptoms Length | 30 days
  Length of COVID-19 associated symptoms from baseline to Day 30 based on self-assessment using daily and weekly symptom diary.
COVID-19 Associated Symptoms Mitigation | 30 days
  Change from baseline through Day 30 of one or more COVID-19 associated symptoms to an improved status
Beck Depression Inventory Score | 0, 8, 14, 30, 60 days
  The Beck Depression Inventory (BDI) is a self-report rating inventory that measures characteristic attitudes and symptoms of depression.
Mental Fatigue Questionnaire Score | 0, 8, 14, 30, 60 days
  Mental Fatigue Questionnaire Score is a self-reported scale that measure mental fatigue.
Pulse Oxygen Saturation | 0, Days 4, 8, 14, 21,30, 60 days
  A Pulse Oxygen Saturation (SpO2) measures how much oxygen is in someone's blood.
Heart Rate Variability by ECG | 0, 8, 14, 60 days
  Change from baseline in Heart Rate Variability by ECG at Days 8, 14, and 60.
Transthoracic echocardiogram | 0, 8, 60 days
  Transthoracic echocardiogram measures of left ventricular function, right ventricular function, and Doppler-derived pulmonary artery pressure.
Frequency of Urgent Care | 0, 30, 60 days
  Number and length of patient's doctor/urgent care/emergency room visit.
C-reactive protein Levels | 0, 8, 14, 21 days
  CRP from serum of blood samples.
D-dimer Levels | 0, 8, 14, 21 days
  D-dimer from serum of blood samples methodology using blood samples
Cytokine Levels | 0, 8, 14, 21 days
  Measure IL-6, TNF-alpha etc from serum of blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Phrsai, Study Director — Proxima
Locations (4):
- United States (4):
  - NewportNativeMD, Newport Beach, California
  - Assuta Family Medical Group, North Hollywood, California
  - Innovation Clinical Trials, Miami, Florida
  - United Memorial Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No